CLINICAL TRIAL: NCT03810287
Title: The Use Of Domperidone For The Relief Of Refractory Upper Gastrointestinal GI Symptoms
Status: No longer available | Type: Expanded Access
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1410014717
Record Dates: First submitted 2018-05-31; First posted 2019-01-18 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Domperidone

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Domperidone — Domperidone will be prescribed for patients with upper GI symptoms at an initial dose of 10 mg up to 4 times a day (prior to each meal and at bedtime). It is possible that the dose of domperidone may be increased to 20 mg if symptoms are not adequately controlled on the initial dose.

SUMMARY:
To prescribe oral domperidone for patients with upper GI symptoms who have failed or suffered adverse effects from standard medical therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to prescribe oral domperidone for patients with upper GI symptoms who have failed or suffered adverse effects from standard medical therapy

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are 18 years of age or older
2. Symptoms or manifestations secondary to Gastro esophageal reflux disease (GERD) (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy.

Exclusion Criteria:

1. i. History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.

   ii. Clinically significant bradycardia, sinus node dysfunction, or heart block.

   iii. Prolonged QTc (QTc>450 milliseconds for males, QTc>470 milliseconds for females)

   iv. Clinically significant electrolyte disorders.
2. Gastrointestinal hemorrhage or obstruction.
3. Presence of a prolactinoma (prolactin-releasing pituitary tumor).
4. Pregnant or breast feedings female.
5. Known allergy to domperidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jill Deutsch, MD, Principal Investigator — Yale University
Locations (1):
- Yale Digestive Diseases, New Haven, Connecticut, United States